CLINICAL TRIAL: NCT03285334
Title: The Effect of 3D Instrumentation Versus Rotary Instrumentation on Postoperative Pain and Bacterial Reduction in Necrotic Oval Canals: A Randomized Clinical Trial
Brief Title: 3D Instrumentation Versus Rotary Instrumentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Sameeh Emara, assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-09-19
Record Dates: First submitted 2017-09-13; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * The patients will drag an envelope and will not know to which group they will be assigned.
  * The patients who already do not know their treatment group will assess the level of their post-operative pain and will record the number of analgesic tablets used.
  * The laboratory technician at the microbiological department will not know the treatment group of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XP-endo Shaper (Experimental): The XP-endo Shaper is an innovative single instrument manufactured from Max wire. Its special ability to shift crystalline structure at body temperature in order to adapt to the root canal wall, has provided a unique instrument with the promise of anatomical shaping.
  Interventions: Device: XP-endo Shaper
- iRace (Active Comparator): rotary files
  Interventions: Device: iRace files

INTERVENTIONS:
Device: XP-endo Shaper — mechanical preparation in a 3D manner using Xp-endo Shaper
  Other Names: anatomical (3D) shaping file
  Arms: XP-endo Shaper
Device: iRace files — rotary mechanical preparation
  Other Names: rotary files
  Arms: iRace

SUMMARY:
enrollment of the patient after diagnosis, radiographic evaluation, and signing the informed consent.

allocation of the patient to either intervention or control group. After anaesthesia and access cavity, the first root canal sample will be taken. Endodontic treatment will be completed in one visit. The second root canal sample will be taken. Patients will be asked to evaluate their postoperative pain level using VAS scale at 6, 12, 24 hours, and daily up to 5 days. Patients will record the number of analgesics if any taken.

DETAILED DESCRIPTION:
After diagnosing the case as asymptomatic pulp necrosis and confirming that the patient conforms to all eligibility criteria, (R.S) will enroll the patient in the study.

the operator will complete treatment of all cases in single visit as following:

1. Anesthetizing the tooth using inferior alveolar nerve block technique
2. Removal of Caries and/or coronal restorations completely with sterile bur and rubber dam will be applied.
3. Preparation of access cavity using another sterile round carbide bur size 3 and Endo-z bur .
4. (R.S) will take the preinstrumentation root canal sample (S1)
5. Confirming the patency of the root canals using stainless steel hand K-files size #10 and #15 . Working length will be determined .
6. In the intervention group, (R.S) will perform mechanical preparation in a 3D manner using Xp-endo Shaper single file in an endodontic motor at a speed of 800 rpm and a torque of 1 Ncm.
7. In the control group, mechanical preparation will be done using rotary iRace files (#25/0.04, #30/0.04, and #40/0.04) at a speed of 600 rpm and a torque of 1.5 Ncm. The canal will be irrigated and recapitulated after the use of each instrument.
8. EDTA gel will be used as a lubricant. The canals will be thoroughly irrigated using 3ml of 2.5% sodium hypochlorite.
9. The canal will then be dried by using sterile paper points and then flushed with 5 ml of 5% sodium thiosulfate to inactivate the NaOCl. The postinstrumentation sample (S2) will be taken from the canals.
10. Master cones will be fitted to the working length and a radiograph will be taken to ensure proper length.
11. (R.S) will complete obturation using AdSeal resin-based root canal sealer .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Adult patients.
2. Age between 20-40 years old.
3. Males & Females.
4. Asymptomatic necrotic mandibular premolars with or without periapical radiolucency.
5. Normal occlusal contact with the opposing teeth.
6. Patients accepting to participate in the study.

Exclusion criteria:

1. Medically compromised patients
2. Pregnant women
3. If analgesics or antibiotics have been administrated by the patient during the past 12 hours preoperatively
4. Patients reporting bruxism or clenching
5. Teeth that shows:

   * Association with acute periapical abscess and swelling
   * Greater than grade I mobility or pocket depth greater than 5mm
   * No restorability

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | up to 5 days
  Degree of postoperative pain will be measured by the patients using modified VAS

SECONDARY OUTCOMES:
intracanal bacterial reduction | 6 hours
  The intra-canal bacterial count will be determined using culture technique in the microbiological department, Cairo University. Samples in RTF vials will be dispersed with vortex for 30 seconds by the laboratory technician. The RTF solution will be serially diluted one-tenth dilution and spiral plated onto the agar medium. The plates will be incubated at 37ₒc aerobically and anaerobically.
  The resultant anaerobic growth will be quantified by evaluating the colony forming units (CFU) on the agar medium under the microscope and the number of CFU per milliliter of each dilution will be calculated for each sample.
Incidence of analgesic intake | up to 5 days
  In case of presence of moderate or severe postoperative pain, (R.S) will instruct the patients to take only one capsule of placebo given to him/her at the end of the visit (Powdered milk packed in opaque capsules)

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Emara, Principal Investigator — faculty of oral and dental medicine - cairo university
Locations (1):
- Faculty of Oral and Dental Medicine - Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No